CLINICAL TRIAL: NCT04004026
Title: The Validity and Reliability of 3 Meter Backwards Walk Test in Multiple Sclerosis Patients
Brief Title: 3 Meter Backwards Walk Test and Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, zekiye ipek katırcı kırmacı, assistant professor, Kahramanmaras Sutcu Imam University
Other Study IDs: SankoU
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis; Walking, Difficulty; Balance; Distorted
Keywords: Multiple Sclerosis; 3-m backwards walk; Balance; Fall risk; validity; reliability
MeSH Terms: conditions — Multiple Sclerosis; Mobility Limitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (1):
- Multiple sclerosis patient: First day, first evaluator will perform all tests, and second day, second evaluator will perform 3 m backwards walk test.
  Interventions: Other: Assesment

INTERVENTIONS:
Other: Assesment — 3-m backwards walk test, timed up and go test, 12-item MS Walking Scale, 2-min walk test, timed 25-foot walk test, 4-square step test.

SUMMARY:
Multiple Sclerosis (MS) is an autoimmune, demyelinating disease of the central nervous system that causes different levels of disability with motor and sensory loss. Although the signs and symptoms of the disease vary according to the location of the lesion; loss of strength, spasticity, sensory disturbances, fatigue, ataxia, autonomic dysfunction and decreased visual acuity are frequently seen. One of the most important causes of loss of function is balance problems. Balance problems, on the other hand, result in falls that cause severe injuries. One of the most important goals in the rehabilitation of individuals with MS is to increase their performance by minimizing the risk of falling in their daily lives. For medical professionals, many medical history questionnaires, self-assessment measures and performance-based tests have been developed to determine the risk of falls. Performance-based functional assessments consist of a timed walk and walk test, functional skill, balance and fall risk, 5 times sit-and-go test and Berg Balance Test, 4 square step test and gait speed measurement tests. These tests include the ability to walk forward and revolve around ones priorities. However, walking is a more difficult activity as it involves neuromuscular control and is dependent on proprioception and protective reflexes. In daily life activities, there is a need to walk backwards to perform tasks such as leaning against a chair and opening the door. This movement can be quite challenging especially for elderly people with neurological deficits. It has been noted that the mechanical measurements of the back support, in particular the speed, the step length, and the double support surface are significantly reduced in older adults. In a study conducted in geriatric individuals, it was shown that walking backward was more sensitive to detect age-related changes in mobility and balance than walking forward. The aim of this study is to determine the validity and reliability of the 3-meter backwards walk test for evaluating performance-based fall risk in individuals with MS.

DETAILED DESCRIPTION:
Gait and mobility are frequently affected functions in MS and have a negative impact on quality of life. Approximately 40% of patients describe walking problems and 70% of individuals in this group are reported to be affected by daily living activities. One of the most important causes of loss of function is balance problems. Balance problems, on the other hand, result in falls that cause severe injuries. One of the most important goals in the rehabilitation of individuals with MS is to increase their performance by minimizing the risk of falling in their daily lives. Therefore, determining the performance-based fall risk of these patients is important in terms of establishing a rehabilitation program and evaluating the treatment results. In this context, researchers have recently reported that assessment of backward gait may be an important clinical tool to determine the risk of falling, especially in individuals with balance problems. However, it has not been investigated whether backward gait is often associated with performance and balance tests in individuals with MS who have balance problems. The aim of this study is to determine the validity and reliability of the 3-meter backwards walk test for evaluating performance-based fall risk in individuals with MS.

ELIGIBILITY:
Inclusion Criteria:

* EDSS score is 4 or less,

Exclusion Criteria:

* Pregnancy or in the first 3 months after birth,
* Corticosteroid treatment in the last month
* Using medication that will affect walking in the last 1 month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Multiple Sclerosis patient
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
3 m backwards walk test | First and second days
  465/5000 A distance of 3 m is measured and marked with black tape. Individuals are asked to follow the heel and black band. With the 'start' command they are asked to walk backwards quickly. When the distance of 3 m is completed, a stop is instructed. Individuals are not allowed to run during the test. They are allowed to look back if they wish. The assessor walks behind individuals throughout the test. The test is repeated 3 times, the averages are recorded

SECONDARY OUTCOMES:
Timed up and go test | First day
  At the beginning of the test, individuals sit in a chair. A distance of 3 m is determined in front of it. With the start command, he gets up from his seat and walks for 3 m and turns around and walks back and sits. With the Start command, the time in seconds until the seat is fully seated. A shorter duration means that functional mobility is good.
12 Items MS Walking Scale | First day
  It is a 12-item questionnaire that questions the effect of gait in MS. The difficulties experienced by individuals during walking activity during the last 2 weeks are questioned. Each item contains 5 points (1; I am not affected at all; 5; I am fully impressed). Low scores indicate better gait disturbance
2 min walk test | First day
  Individuals are asked to walk as fast as possible without running in a 25 m corridor. The distance they walk for 2 minutes is recorded.
25 foot walk test | First day
  It is an evaluation to evaluate mobility and leg functions. Individuals are asked to walk safely on a flat surface at the highest speed of 7.62 m. Individuals are allowed to use walking aids if necessary. Individuals are asked to walk 3 times. The average of the times is recorded.
4 square step test | First day
  It aims to evaluate dynamic balance and to step forward, sideways and backwards of objects. The square drawn on the floor is divided into 4 equal parts. The number 1 is written in the lower right corner, up to 4 clockwise. With the Start command, individuals are asked to press on the numbers respectively. It is first asked to take a step forward (number 1 and 2) then left (number 3), then backward (number 4). It is then asked to take steps 4 through 1 again. The time is saved.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Ph.D(c), Principal Investigator — Sanko University
Locations (1):
- SANKO University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Carter V, Jain T, James J, Cornwall M, Aldrich A, de Heer HD. The 3-m Backwards Walk and Retrospective Falls: Diagnostic Accuracy of a Novel Clinical Measure. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):249-255. doi: 10.1519/JPT.0000000000000149. PMID 29095771
- See also: The 3-m Backwards Walk and Retrospective Falls: Diagnostic Accuracy of a Novel Clinical Measure. — http://www.ncbi.nlm.nih.gov/pubmed/29095771